CLINICAL TRIAL: NCT06397924
Title: Edible Insects: Good for the Gut and the Globe
Acronym: GGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Tiffany Weir, Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2973
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; Cricket; Chitin; gut microbiome; gut health
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: One group will be given the small chocolate patties containing the insect chitin for 30 days, and the other group will be given the patties containing the placebo. The study was double-blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chitin Fiber (Active Comparator): Chitin Fiber
  Interventions: Dietary Supplement: Chitin Fiber
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Chitin Fiber — Dietary fiber isolated from an edible insect (chitin)
  Arms: Chitin Fiber
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
Edible insects have been eaten by people throughout human history and are consumed today across the globe. Insects are also currently being incorporated into a number of food products in the United States, Canada, and Europe due to their unique nutritional and sustainability attributes. Insects have been touted as an environmental alternative to conventional meat products, but they are unique in containing dietary fiber. The investigators have recently demonstrated in a population of healthy individuals that two weeks of consuming 25 g/day cricket powder may be associated with prebiotic effects by stimulating the growth of Bifidobacterium in the gut. In addition, participants had reduced inflammatory markers in the blood after the cricket intervention. Crickets and other edible insects contain a unique form of fiber called chitin. They would like to explore whether chitin may be responsible for these previously observed effects and particularly if chitin consumption can mitigate symptoms and inflammation associated with the gastrointestinal disorder Irritable Bowel Syndrome (IBS). This project aims to examine the impact of consuming 4 grams of cricket-derived chitin daily for 30 days on the gut microbiota, intestinal and systemic markers of inflammation, and symptom severity and quality of life in individuals with IBS.

DETAILED DESCRIPTION:
The study will take place in the Food and Nutrition Clinical Research Laboratory (FNCRL) located in the Gifford Building Room 216 on the Colorado State University campus. The time commitment for the study is approximately two and a half months, during which participants will spend ~1 hour (15-20 min/visit) at clinic appointments, eat small chocolate bars containing either the cricket chitin or a maltodextrin placebo daily for 30 days each, and collect four stool and four blood samples. (The two-and-a-half-month study will be broken into three parts: one 30-day fiber consumption period, one 14-day break, and a 30-day placebo consumption period.). The participant will be randomly assigned to Group A or Group B, but the treatment schedule for each is the same. One group will be given the small chocolate patties containing the insect chitin for 30 days, and the other group will be given the patties containing the placebo. However, neither the participant nor the research personnel will know whether participants are consuming the placebo or the treatment bars during a specific period until after the study is complete and all data is analyzed.

One group will eat insect fiber-filled chocolate patty for 30 days and then take at least a 14-day break (called a wash-out), followed by 30 days of eating the placebo bars. The other group will eat the placebo patties for 30 days and then take a break of at least 14 days (wash-out), followed by 30 days of eating the cricket fiber patties. During the treatment periods, the participant will consume either 4g of cricket fiber or 4g of maltodextrin (a type of sugar) included in the chocolate patties.

At the baseline visits, as well as at the end of each treatment period, fasted blood and stool samples will be collected by trained research personnel at the FNCRL. This means that participants will have a total of four (4) clinic visits during the study. The participant will be required to drop off the first stool sample at a specified location after the first visit. Subsequent stool kits will be returned at the scheduled clinic visit. Additionally, at each visit, the participant will be weighed, and hip and waist circumference will be measured. The participant will also fill out several forms, including questionnaires about any IBS-related symptoms and about their quality of life. Finally, the participant will take home a form to track their daily bowel movements and a 3-day diet diary to record what the participant eats at the beginning and end of each treatment period.

All blood samples will be collected at Colorado State University by a trained professional. The research team will provide the participant with collection materials and instructions, and the participant will perform fecal sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older with a medical diagnosis of Irritable Bowel Syndrome (IBS) and/or recurrent abdominal pain greater than 1 time per week persistent for at least 3 months while also meeting 2 of the 3 criteria for IBS diagnosis according to the Rome IV assessment. Both adult males and females of any race or ethnicity will be included in this study. (Rome IV Diagnostic Criteria for IBS link: www.mdcalcl.com/rome-iv-diagnostic-criteria-irritable-bowel-syndrome-ibs)

Exclusion Criteria:

* pregnant and lactating women,
* individuals taking antibiotics or who have recently taken antibiotics (within 60 days of the study start date),
* individuals with any self-reported shellfish, milk, or soy allergies
* individuals with a current diagnosis of inflammatory bowel disease, gastrointestinal cancers, other cancers, liver or kidney disease,
* individuals reporting current medication and dietary supplement use, along with the presence of other metabolic diseases, will be assessed on a case-by-case basis and may result in study exclusion
* individuals who feel that they will not be able to adhere to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Examine the impact that consuming 4 grams of cricket-derived chitin daily for 30 days has on the gut microbiota, intestinal and systemic markers of inflammation, and symptom severity and quality of life in individuals with IBS. | The time commitment for the study is approximately two and a half months, during which participants will spend ~1 hour (15-20 min/visit) at clinic appointments, eat small chocolate bars containing either the cricket chitin or a maltodextrin placebo daily

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Weir, MSc,PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Stull VJ, Finer E, Bergmans RS, Febvre HP, Longhurst C, Manter DK, Patz JA, Weir TL. Impact of Edible Cricket Consumption on Gut Microbiota in Healthy Adults, a Double-blind, Randomized Crossover Trial. Sci Rep. 2018 Jul 17;8(1):10762. doi: 10.1038/s41598-018-29032-2. PMID 30018370
- [Background] FAO, IFAD, UNICEF, WFP & WHO. The State of Food Security and Nutrition in the World 2018. Building Climate Resilience for Food Security and Nutrition. (2018).
- [Background] Korpe PS, Petri WA Jr. Environmental enteropathy: critical implications of a poorly understood condition. Trends Mol Med. 2012 Jun;18(6):328-36. doi: 10.1016/j.molmed.2012.04.007. Epub 2012 May 25. PMID 22633998
- [Background] Prendergast A, Kelly P. Enteropathies in the developing world: neglected effects on global health. Am J Trop Med Hyg. 2012 May;86(5):756-63. doi: 10.4269/ajtmh.2012.11-0743. PMID 22556071
- [Derived] Vita AA, Teo S, Murphy C, Khandaker AM, Hart RA, Mathews P, Wilson JW, Chaparro J, Aquilino T, Dinsmore I, Wei Y, Stull VJ, Weir TL. Safety, tolerability, and preliminary effects of cricket chitin for adults with IBS: a double-blind randomized crossover pilot trial. Food Funct. 2025 Sep 15;16(18):7434-7454. doi: 10.1039/d5fo01540e. PMID 40891151